CLINICAL TRIAL: NCT00726765
Title: Observational Trial on the Value of Diagnostic Criteria in the Diagnosis of Spinal Spondyloarthropathies in Patients With Chronic Low Back Pain
Brief Title: Diagnostic Criteria in the Diagnosis of Spinal Spondyloarthropathies in Patients With Chronic Low Back Pain (Study P05320)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05320
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Spinal Spondyloarthropathies; Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Referral Strategy 1: Patient meets at least one of the following three criteria:
  1. Inflammatory back pain
  2. Human leukocyte antigen B27 (HLA-B27)
  3. Sacroiliitis demonstrated by imaging (X-ray, magnetic resonance imagining [MRI], bone scan [if previously available])
- Referral Strategy 2: Patient meets at least two of the following six criteria:
  1. Inflammatory back pain
  2. HLA-B27
  3. Sacroiliitis (on imaging)
  4. Family history of AS
  5. Good response of back pain to nonsteroidal anti-inflammatory drugs (NSAIDs)
  6. Known Extra Articular Manifestations (Uveitis, Iridocyclitis, Psoriasis, Inflammatory Bowel Disease)

SUMMARY:
This is a multi-national, multi-site, observational study to determine which of two strategies, when used by referring physicians is superior in the diagnosis of axial spondyloarthritis (AS) by rheumatologists.

DETAILED DESCRIPTION:
Subjects will be selected using a non-probability sampling method. For each center of excellence, the local network of referring physicians will be assigned, according to a random code in a 1:1 ratio, to use one of the two referral strategies for eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* A subject must have back pain of unknown origin, of more than 3 months' duration, and with onset before age 45.
* A subject must be willing to give written informed consent and be able to adhere to visit schedules.

Exclusion Criteria:

* Established diagnosis of spondyloarthropathies at the time of referral.
* Any clinically significant condition or situation, other than the condition being studied, that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each of several participating national centers of excellence will establish a network with local primary care physicians or their equivalent who will work with the center of excellence and will provide referrals of suitable patients.
Sampling Method: Non-Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine which of two referral strategies, when used by referring physicians, is superior in the diagnosis of AS by rheumatologists. | Approximately 3-6 months

SECONDARY OUTCOMES:
To determine which of the referral criteria proposed, or which combination of referral criteria, is the most successful and workable in the diagnosis of AS when used by referring physicians. | Approximately 3-6 months
To describe the demographics and disease characteristics of patients diagnosed with AS. | Approximately 3-6 months
To compare patient-derived data with physician data to determine whether the former alone can serve as effective screening for AS. | Approximately 3-6 months

REFERENCES:
- [Background] Sieper J, Srinivasan S, Zamani O, Mielants H, Choquette D, Pavelka K, Loft AG, Geher P, Danda D, Reitblat T, Cantini F, Ancuta C, Erdes S, Raffayova H, Keat A, Gaston JS, Praprotnik S, Vastesaeger N. Comparison of two referral strategies for diagnosis of axial spondyloarthritis: the Recognising and Diagnosing Ankylosing Spondylitis Reliably (RADAR) study. Ann Rheum Dis. 2013 Oct;72(10):1621-7. doi: 10.1136/annrheumdis-2012-201777. Epub 2012 Oct 13. PMID 23065731